CLINICAL TRIAL: NCT06547684
Title: Effects of Focused Extracorporeal Shock Wave Therapy on Spastic Equinus Foot in Stroke Patients: a Randomized Controlled Trial
Brief Title: Extracorporeal Shock Wave Therapy on Spastic Equinus Foot in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teresa Mateu Campos (Other)
Responsible Party: Sponsor-Investigator, Teresa Mateu Campos, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-OCF-2019-02
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Equinus Deformity; Spasticity, Muscle
Keywords: Stroke; Equinus Deformity; Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Stroke; Equinus Deformity; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Active Comparator): 1 session of fESWT
  Interventions: Device: fESWT
- GROUP 2 (Experimental): 3 sessions of fESWT (1 session per week for 3 consecutive weeks)
  Interventions: Device: fESWT

INTERVENTIONS:
Device: fESWT — Shock wave therapy will be applied with Duolith SD1 device (Storz Medical, Tagerwilen, Switzerland). Therapy will be administered in the gastrocnemius medial and lateral and in the soleus muscles.
  Parameters: 0.15mJ/mm2, 4-5 Hz, 1500 shoots/muscle.

SUMMARY:
The goal of this study is to evaluate long term effects of focused extracorporeal shock wave therapy (fESWT) on triceps surae spasticity in stroke patients according to the number of sessions applied.

Hypothesis: 3 sessions of fESWT on equinus foot in stroke patients improve spasticity and functionality for longer term than 1 session of fESWT.

DETAILED DESCRIPTION:
Spasticity is a common complication as a consequence of suffering a stroke and one of the most important causes of disability in this pathology.

Global data estimate that 12 million people world-wide suffer from spasticity of the upper or lower limb. Equinus foot is the most common pattern of the lower extremities.

Previous studies have reported that extracorporeal shock wave therapy (ESWT) is a safe and noninvasive alternative treatment for spasticity.

Although the authors have shown a beneficial clinical effect of the ESWT, outcomes and duration of effect varied across studies.

This is a prospective randomized controlled trial. 60 stroke patients with spastic equinus foot post stroke will enroll in this study.

The participants will be randomly divided into two groups. The first group (control group) will receive 1 session of fESWT, while the second group (experimental group) will receive 3 sessions of fESWT, once a week, for 3 consecutive weeks.

Therapy will be administered directly to the muscle bellies of the gastrocnemius medial and lateral and soleus. The muscle belly will be located by ultrasonography.

The primary outcome is modified Ashworth scale. Secondary outcomes are passive range of ankle motion, mobility and balance test, spasm frequency scale and quality of life scales.

Participants will be evaluated by the same researcher before the first shock wave therapy and after the last session of fESWT will be done periodic revisions on weeks 1, 4, 8, 12, 20, 24, 36 and 48. Adverse events will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Time from stroke (ischemic o hemorrhagic) onset of at least 6 months
* Spastic equinus foot: triceps surae tone grade at least 1+ on the MAS score
* Ability to walk alone with or without aids

Exclusion Criteria:

* Fixed ankle joint contracture
* Severe medical problems
* Treatment of the affected leg with botulinum toxin in the las 6 months
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  A manual measurement of the resistance os muscles during passive stretching. Score from 0 to 4, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Passive Ankle range of motion (PROM) | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Measure with goniometer
Visual Analogue Scale (VAS) Pain Score | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Pain Score: from 0 (no pain) to 10 (the worst imaginable pain)
10 Meters Walk Test | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Measure the gait speed
Test Up and Go (TUG) | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Asses the mobility and balance
Spasm Frequency Scale | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Estimate muscle spams. Score 0 (no spams) to 4 (>10 spams)
Test 6 Minutes Walking | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Asses walking resistance
Fall Skip Device | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  Assesment of fall risk
Stroke Quality of Life Scale (ECVI-38) | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  A questionnaire of 38 items: from 1 (no problem) to 190 (the worst situation)
Self Report Spasticity Scale (SRSS) | Before the first shock wave therapy and 1,4,8,12,20,24,36 and 48 weeks after the last session of ESWT.
  A questionnaire of 8 items: from 0 (nothing) to 24 (cpmpletely)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Mª Mateu Campos, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Hospital de la Plana, Vila-real, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo P, Gao F, Zhao T, Sun W, Wang B, Li Z. Positive Effects of Extracorporeal Shock Wave Therapy on Spasticity in Poststroke Patients: A Meta-Analysis. J Stroke Cerebrovasc Dis. 2017 Nov;26(11):2470-2476. doi: 10.1016/j.jstrokecerebrovasdis.2017.08.019. Epub 2017 Sep 13. PMID 28918085
- [Background] Lee JY, Kim SN, Lee IS, Jung H, Lee KS, Koh SE. Effects of Extracorporeal Shock Wave Therapy on Spasticity in Patients after Brain Injury: A Meta-analysis. J Phys Ther Sci. 2014 Oct;26(10):1641-7. doi: 10.1589/jpts.26.1641. Epub 2014 Oct 28. PMID 25364134
- [Background] Taheri P, Vahdatpour B, Mellat M, Ashtari F, Akbari M. Effect of Extracorporeal Shock Wave Therapy on Lower Limb Spasticity in Stroke Patients. Arch Iran Med. 2017 Jun;20(6):338-343. PMID 28646841